CLINICAL TRIAL: NCT05592886
Title: A Multicenter, Double Blinded Randomized Controlled Trial of a Novel Oral Synbiotic Formula in Reducing Advanced Adenoma Recurrence and Colorectal Neoplasia-related Bacterial Gene Markers
Brief Title: A Novel Oral Synbiotic Formula in Reducing Advanced Adenoma Recurrence and Colorectal Neoplasia-related Bacterial Gene Markers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Inner Mongolia People's Hospital (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022.360
Record Dates: First submitted 2022-10-17; First posted 2022-10-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Neoplasms; Colorectal Adenoma; Colorectal Cancer; Advanced Adenoma
Keywords: Adenoma recurrence; Bacterial marker
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Receive SMT04 formula
  Interventions: Other: SMT04 formula
- Placebo arm (Placebo Comparator): Receive active placebo
  Interventions: Other: Active placebo

INTERVENTIONS:
Other: SMT04 formula — The SMT04 formula is a synbiotic containing probiotics and prebiotics
  Arms: Intervention arm
Other: Active placebo — The active placebo is 2 mg Vitamin C with an inert substance made of starch filler. The flavor, coloring and appearance are unidentifiable to the study product.
  Arms: Placebo arm

SUMMARY:
This multicenter, double blinded randomized controlled trial aims to assess the efficacy of a novel oral synbiotic formula (SMT04) in reducing advanced adenoma recurrence and colorectal neoplasia-related bacterial gene markers after endoscopic resection of colorectal advanced neoplasia.

DETAILED DESCRIPTION:
Recent evidence has demonstrated the association between altered gut microbiome environment and the progression of colorectal cancer (CRC) from its precancerous lesions. Some pathogenic species of bacteria, including Fusobacterium nucleatum, Escherichia Coli and Bacteroides fragilis, have shown to be significantly enriched in CRC patients. This gut dysbiosis process also brings with its diagnostic potential for recurrent adenomas. Previous study found a panel of bacterial gene markers, including "m3" from Lachnoclostridium, F. nucleatum (Fn), Bacteroides clarus (Bc) and Clostridium hathewayi (Ch) could be used in detecting adenoma recurrence after polypectomy in a retrospective study. In addition, these microbial biomarkers may have prognostic potential and provide an option as therapeutic target.

Probiotics, including the genera Bifidobacterium and Lactobacillus, have shown to be able to inhibit tumorigenesis and progression of CRC in animal studies. Prebiotics are non-digestible dietary ingredients with protective effects against cancer by selectively stimulating the growth and activity of beneficial colonic microbiota. The combination of probiotics and prebiotics, known as synbiotic, may be more efficient in preventing CRC than either one alone.

The investigators' unpublished data showed that the new probiotic formula containing Bifidobacterium strains has a negative correlation with CRC-related bacterial gene markers. Subjects treated with SMT04 showed significantly higher levels of the individual Bifidobacterium species at week 2 to week 5 compared with baseline levels. There was a significant decrease in the bacterial gene markers (Fn, m3 and 4Bac CRC risk score) from week 2 to week 12 compared with baseline levels in the SMT04 group but not in the control group. The synbiotic formula (SMT04) is the combination of probiotic formula and several heat-resistant prebiotics. It remains unclear that whether this synbiotic formula can produce a sustained effect in reduction of advanced adenoma recurrence and colorectal neoplasia related bacterial gene markers in long-term.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have advanced colorectal neoplasia* removed and confirmed by histopathology;
* They have received high quality colonoscopies before or during endoscopic resection (defined as a full colonoscopy with successful caecal intubation, and a Boston Bowel Preparation Scale ≧2 in each colonic segment) with no residual colorectal neoplasia;
* Aged 18-90 years old;
* Written informed consent obtained

  * An advanced colorectal neoplasia is defined as an advanced adenoma, sessile serrated lesion or non-invasive colorectal cancer (stage Tis or T1a). Advanced adenoma is defined as an adenoma larger than 10mm, and/or with villous component ≥20%, and/or harboring high grade dysplasia.

Exclusion Criteria:

* Known residual colorectal neoplasia not removed (except hyperplastic polyps);
* Contraindications to endoscopic resection due to deep submucosal invasion (stage T1b or above);
* Prior surgical resection of colon;
* Personal history of hereditary polyposis syndrome or inflammatory bowel disease;
* Known pregnancy or lactation;
* Immunocompromised status (e.g. on immunosuppressants (except 5-aminosalicylic acid or short term use of corticosteroids <4 weeks), on chemotherapy, bone marrow or solid organ transplant, human immunodeficiency virus, congenital immune deficiency);
* Advanced comorbid conditions (defined as American Society of Anesthesiologists grade 4 or above);
* Refusal to undergo surveillance colonoscopy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 649 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of metachronous recurrent advanced colorectal neoplasia at year 1 (local or at other sites). | 1 year
  The proportion of patients with metachronous recurrent advanced neoplasia at year 1

SECONDARY OUTCOMES:
Incidence of recurrent colorectal adenomas at year 1 | 1 year
  The proportion of patients with metachronous recurrent adenoma at year 1
Number of recurrent advanced neoplasia at year 1 | 1 year
  The number of recurrent colorectal advanced neoplasia per patient both in intervention and placebo arm
Number of recurrent adenomas at year 1 | 1 year
  The number of recurrent colorectal adenoma per patient both in intervention and placebo arm
Changes in the levels of bacterial gene markers | 1 year
  The change in the level of four bacterial gene markers and combined risk score tested by qPCR
Correlation between recurrent advanced colorectal neoplasia and the changes in levels of bacterial gene markers | 1 year
  Correlation of incidence rate of recurrent advanced colorectal neoplasia and the changes in the level of four bacterial gene markers and combined risk score tested by qPCR
Correlation between recurrent adenoma and the changes in levels of bacterial gene markers | 1 year
  Correlation of incidence rate of recurrent adenoma and the changes in the level of four bacterial gene markers and combined risk score tested by qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Louis Lau, Principal Investigator — Prince of Wales Hospital
Locations (2):
- Inner Mongolia People's Hospital, Hohhot, Inner Mongolia, China
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No